CLINICAL TRIAL: NCT00862511
Title: A Prospective Randomized Comparison of Serum Metal Ion Levels After Implantation of Coated and Uncoated Knee Prostheses
Brief Title: Serum Metal Ion Concentration After Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KneeIon
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthritis; Metal Ion Levels
Keywords: metal ion concentration; total knee arthroplasty; metal hypersensitivity
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coated Total Knee Arthroplasty (Experimental): allergy coated TKA
  Interventions: Device: Coated Total Knee Arthroplasty
- Standard Total Knee Arthroplasty (Active Comparator): normal TKA
  Interventions: Device: Standard Total Knee Arthroplasty

INTERVENTIONS:
Device: Coated Total Knee Arthroplasty — Implantation of a coated Total Knee Arthroplasty
  Arms: Coated Total Knee Arthroplasty
Device: Standard Total Knee Arthroplasty — Implantation of a Standard Total Knee Arthroplasty
  Arms: Standard Total Knee Arthroplasty

SUMMARY:
All metal implants release metal ions because of corrosion. Total knee arthroplasty implants have large metal surface areas and therefore substantial potential for corrosion. It is planned to compare changes in serum levels of metal ions in patients after implantation of cemented unconstrained total knee arthroplasty covered with or without a passivating surface. Serum concentrations of chromium, cobalt, molybdenum and nickel will be analyzed and compared between the two groups, as well as with those of 130 control patients without implants.

ELIGIBILITY:
Inclusion Criteria:

* Indication for TKA in primary oder secondary osteoarthritis of the knee
* Patient's consent

Exclusion Criteria:

* Additional Implants present
* Allergy against constituents of implant or cement
* Any malignancies
* Renal insufficiency
* Any additional serious disease complicating the participation in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Metal ion concentration in serum after TKA (Cr, Co, Mb, Ni) | 1 y and 5y

SECONDARY OUTCOMES:
Hypersensitivity against metal | 1 y

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, MD, Principal Investigator — University Hospital Dresden, Orthopaedic Department; Stephan Kirschner, MD, Principal Investigator — University Hospital Dresden, Orthopaedic Department
Locations (1):
- University Hospital Dresden, Orthopaedic Department, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lutzner J, Beyer F, Lutzner C, Thomas P, Summer B. Increased inflammatory response is associated with less favorable functional results 5 years after total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2023 Apr;31(4):1316-1322. doi: 10.1007/s00167-021-06836-w. Epub 2022 Feb 11. PMID 35147719
- [Derived] Lutzner J, Dinnebier G, Hartmann A, Gunther KP, Kirschner S. Study rationale and protocol: prospective randomized comparison of metal ion concentrations in the patient's plasma after implantation of coated and uncoated total knee prostheses. BMC Musculoskelet Disord. 2009 Oct 14;10:128. doi: 10.1186/1471-2474-10-128. PMID 19828019